CLINICAL TRIAL: NCT00198055
Title: An Open-Label Study of Aripiprazole in Children and Adolescents With Autistic Disorder
Brief Title: A Study of Aripiprazole in Children and Adolescents With Aspergers and Pervasive Developmental Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0302-24
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Asperger's Disorder; Pervasive Developmental Disorder
Keywords: Aggression; Behavioral symptoms
MeSH Terms: conditions — Asperger Syndrome; Child Development Disorders, Pervasive; Aggression; Behavioral Symptoms | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aripiprazole (Experimental): Aripiprazole 5 mg per day for 2 weeks, then can be increased to 10mg per day if tolerated for 2 weeks, then can be increased to 15 mg per day for 4 weeks.
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: aripiprazole — Aripiprazole 5 mg per day for 2 weeks, then can be increased to 10mg per day if tolerated for 2 weeks, then can be increased to 15 mg per day for 4 weeks.
  Other Names: Abilify

SUMMARY:
The purpose of this study is to develop a better tolerated and more effective pharmacologic treatment for individuals with Asperger's Disorder and Pervasive Developmental Disorder. This is an open-label investigation of aripiprazole in the management of the maladaptive behaviors of autistic disorder. We hypothesize that aripiprazole will be effective for reducing aggression and repetitive behavior.

DETAILED DESCRIPTION:
Pervasive developmental disorders (PDD) are characterized be severe impairments in social interaction and communication in addition to restricted patterns of interests and activities. Research suggests that a dysregulation of the dopamine and serotonin systems contributes to these interfering behaviors in individuals with PDD. After benefits of typical neuroleptics were reported in subjects with PDD's, research shifted to the atypical antipsychotics, which have been shown to be better tolerated and effective in this population. However, the atypical antipsychotics have also been associated with adverse effects. Thus there remains a need for a novel pharmacotherapy that would be safe and effective for children and adolescents with PDD's including Asperger's disorder and PDD Not Otherwise Specified (PDD NOS). We hypothesize that aripiprazole will be effective for reducing aggression and repetitive behavior. We also hypothesize that aripiprazole will be well tolerated, with low risk for extrapyramidal symptoms, hyperprolactinemia, weight gain, or corrected QT interval (QTc) prolongation. In addition, this open-label study will serve to stimulate more definitive, controlled research.

ELIGIBILITY:
Inclusion Criteria:

* Mental age of 18 months
* Diagnosis of Asperger's Disorder or Pervasive Developmental Disorder
* Good health overall
* Free of all psychotropic medication for 2 weeks

Exclusion Criteria:

* Weight less than 15kg
* Subjects who have received an adequate trial of aripiprazole
* An active seizure disorder
* A significant medical condition
* History of neuroleptic malignant syndrome
* Females with positive Beta human chorionic gonadotropin(HCG) pregnancy test

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The Clinical Global Impression(CGI)Improvement Scale. | Every 2 Weeks
The Irritability subscale of the Aberrant Behavior Checklist (ABC) | Every 2 weeks

SECONDARY OUTCOMES:
The Clinical Global Impression Severity Scale. | At baseline and endpoint
The Compulsion subscale of the Children's Yale-Brown Obsessive-Compulsive(CY-BOCS). | At baseline and endpoint
The Vineland Maladaptive Behavior Subscale. | At baseline and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A. Stigler, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital, Riley Child and Adolescent Psychiatry Clinic, Indianapolis, Indiana, United States